CLINICAL TRIAL: NCT00741247
Title: Minimally Invasive Mediastinal Staging of Potentially Operable Lung Cancer With Endobronchial Ultrasound Guided Transbronchial Needle Aspiration(EBUS-TBNA) and Transesophageal Aspiration Using Ultrasonic Bronchoscope (EUS-B-FNA)
Brief Title: Mediastinal Staging of Lung Cancer With EBUS-TBNA and EUS-B-FNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: National Cancer Center, Korea, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCCCTS-08-332
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Lung Cancer
Keywords: staging; Endobronchial ultrasound; Endoscopic ultrasound
MeSH Terms: conditions — Lung Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Bronchoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: EBUS-TBNA, EUS-B-FNA (EUS-FNA with bronchoscope) — EBUS-TBNA is a bronchoscopic diagnostic method that enables real time aspiration of paratracheal and peribronchial lesions. EUS-FNA is a procedure to obtain samples through the esophagus under real-time ultrasound guidance. In this study, EUS-FNA will be applied using a ultrasonic bronchoscope (EUS-B-FNA).

SUMMARY:
The purpose of this study is to find a role of EUS-B-FNA in the mediastinal staging of potentially operable lung cancer. The investigators perform EBUS-TBNA and EUS-B-FNA on potentially operable lung cancer patients. The investigators perform EBUS(+/- TBNA) and EUS-B (ultrasonographic examination through the esophagus) on all subjects. EUS-B-FNA will be performed on inaccessible nodes or difficult nodes to be sampled by EBUS-TBNA. Additional diagnostic values of EUS-B-FNA as compared to EBUS-TBNA alone will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed or strongly suspected potentially operable non-small cell lung cancer (NSCLC)
* Potentially operable patients

Exclusion Criteria:

After staging work-up for NSCLC, including bronchoscopy,CT of the chest and upper abdomen, integrated PET/CT and brain MRI (and/or bone scan)

* M1 disease
* Inoperable T4 disease
* Mediastinal infiltration or extranodal invasion of the mediastinal lymph node visible on chest CT.
* Confirmed supraclavicular lymph node metastasis
* Pancoast tumors
* Medically inoperable patients
* Contraindications for bronchoscopy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The diagnostic values of EBUS-TBNA plus EUS-B-FNA as compared to EBUS-TBNA alone | June 2009

SECONDARY OUTCOMES:
The Proportion and the location of lymph nodes accessible by EBUS-TBNA and EUS-B-FNA. | June 2009

CONTACTS AND LOCATIONS:
Locations (1):
- NCCKorea, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Hwangbo B, Lee GK, Lee HS, Lim KY, Lee SH, Kim HY, Lee HS, Kim MS, Lee JM, Nam BH, Zo JI. Transbronchial and transesophageal fine-needle aspiration using an ultrasound bronchoscope in mediastinal staging of potentially operable lung cancer. Chest. 2010 Oct;138(4):795-802. doi: 10.1378/chest.09-2100. Epub 2010 Mar 26. PMID 20348194